CLINICAL TRIAL: NCT02707133
Title: Validation of a Virtual Clinic for Choroidal Nevomelanocytic Lesions: Safety, Patient Acceptability and Health Economics Analysis
Brief Title: Validation of a Virtual Model of Service Delivery for Choroidal Nevi
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: Nevus Protocol v1.0
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Choroidal Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Choroidal nevomelanocytic lesions have a high prevalence affecting up to 7% of the entire population and are increasingly incidentally identified during routine eye check- ups in community optometry services. Given the tendency to err on the side of caution, there is evidence of excessive referrals challenging service delivery in both tertiary eye units and specialist ocular oncology services. Although previous studies have examined the natural history and risk factors for growth of choroidal nevomelanocytic lesions, optimal delivery of management remains uncertain. Management approaches display diversity with respect to the number and type of baseline investigations, the duration and frequency of monitoring of relevant patients. Utilisation of the skills of allied health professionals in appropriate cases would allow streamlining service delivery in a socialised healthcare system, maximise capacity, and allow community services to play an enhanced role. However, the evidence for this model of delivery is lacking. Within existing models of care for these lesions, patients are faced with delays, need for more than one attendances to the hospital and increased anxiety around prognosis.

This project aims to answer the question of whether these low-risk, bland incidental findings might possibly be managed by allied health professionals with the use of clinical imaging and specific algorithms to make appropriate management decisions. We aim to validate a model of service delivery on a virtual basis that will accommodate for capacity pressures to accept all relevant referrals, while offering a safe service and optimising patient experience of care. We will thus validate the setting up of a virtual choroidal nevomelanocytic clinic in terms of safety and patient acceptability. More specifically, the degree of agreement between management decisions made by non-medical graders on the basis of imaging data alone as opposed to gold standard decisions (clinical and imaging tests combined) is examined. Health economics analysis of the proposed service delivery model will be undertaken to demonstrate cost-effectiveness.

ELIGIBILITY:
All patients attending the CNL clinics of MREH/MEH who have offered informed consent will be included in the study. Patients who are then diagnosed with alternate pathologies other than CNL (erroneous referrals) will be excluded from agreement analysis. Recognition of alternate pathologies by non-medical graders will, however, be an additional outcome measure for this project. Cases of Congenital Hypertrophy of the Retinal Pigment Epithelium (CHRPE) will be classified as 'alternate pathology' for the purposes of this study. Exclusion criteria will be media opacities (cornea, lens, vitreous body) precluding adequate visualisation of fundus and incomplete set of imaging data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of MREH and MEH for ocular nevomelanocytic lesions (CNL) will be recruited prospectively into the study.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Degree of agreement (kappa co-efficient) between management decisions reached clinically as opposed to those reached on the basis of imaging tests alone (virtual model) | 18 months
  Validation of the virtual model of service delivery will be sought by calculating the degree of agreement (kappa co-efficient) between management decisions (Discharge, Review or Refer patients) reached by direct clinical examination as opposed to decisions reached through assessing imaging tests only.

IPD SHARING:
Plan to Share IPD: No